CLINICAL TRIAL: NCT00324467
Title: Phase II Trial Investigating Tailoring First-Line Therapy For Advanced Stage Diffuse Large B-Cell Non-Hodgkin's Lymphoma Based on Mid-Treatment Positron Emission Tomography (PET) Scan Results
Brief Title: Tailoring Treatment for B Cell Non-hodgkin's Lymphoma Based on PET Scan Results Mid Treatment
Acronym: LYTPET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H06-00017
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Lymphoma, Non-Hodgkin; Advanced Stage Diffuse Large B-Cell Non-Hodgkin's Lymphoma
Keywords: NON-HODGKIN'S LYMPHOMA; POSITRON EMISSION TOMOGRAPHY; PET; DLBCL; R-CHOP; R-ICE
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Ondansetron; Dexamethasone; Calcium Dobesilate; Diphenhydramine; Acetaminophen; Ifosfamide; Mesna; Carboplatin; Etoposide; etoposide phosphate; Rituximab; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- R-CHOP (Negative Mid-Treatment PET Scan) (Active Comparator): All participants will receive 4 cycles of standard dose R-CHOP chemotherapy administered at 3-weekly intervals. Non-progressing participants will undergo a mid-treatment PET scan along with routine restaging investigations after 4 cycles of R-CHOP. Patients with a negative mid-treatment PET scan (no evidence of abnormal 18F-FDG uptake) will complete therapy with two additional cycles of R-CHOP for a total of 6 cycles of chemotherapy. Patients with a mid-treatment PET scan interpreted to be "indeterminate" or "equivocal" will be recorded as such, but should be considered negative for the purpose of treatment planning and should not prompt a change in therapy.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Ondansetron; Drug: Dexamethasone; Drug: Diphenhydramine; Drug: Acetaminophen; Other: PET Scan
- R-ICE (Positive Mid-Treatment PET Scan (Active Comparator): All participants will receive 4 cycles of standard dose R-CHOP chemotherapy administered at 3-weekly intervals. Non-progressing participants will undergo a mid-treatment PET scan along with routine restaging investigations after 4 cycles of R-CHOP. Patients with a mid-treatment PET scan (abnormal 18F-FDG uptake) will be switched to R-ICE chemotherapy and receive 4 cycles of R-ICE for a total of 8 cycles of chemotherapy.
  Following completion of R-ICE chemotherapy, patients will undergo a post-treatment PET scan along with routine restaging investigations. The post-treatment PET scan will be performed between days 28 and 35 following the final cycle of R-ICE. Patients with a negative post-treatment PET scan will undergo no further therapy. Patients with a positive post-treatment PET scan corresponding to persistent abnormalities on CT scan will be considered for radiation therapy to PET positive sites.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Ondansetron; Drug: Dexamethasone; Drug: Diphenhydramine; Drug: Acetaminophen; Drug: Ifosfamide; Drug: Mesna (IV); Drug: Mesna (oral); Drug: Carboplatin; Drug: Etoposide; Drug: Rituximab; Other: PET Scan

INTERVENTIONS:
Drug: Cyclophosphamide — Dose: 750 mg/m^2 Administration: IV infusion day 1 over 20-60 minutes Schedule: Cycle 1, 2, 3, 4, 5*, 6* (Week 1, 4, 7, 10, 14, 17)
  * Cycles 5 and 6 of R-CHOP will be administered only to patients with a negative mid-treatment PET scan
  Other Names: Cytoxan®, Neosar®
Drug: Doxorubicin — Dose: 50 mg/m^2 Administration: IV Push day 1 Schedule: Cycle 1, 2, 3, 4, 5*, 6* (Week 1, 4, 7, 10, 14, 17)
  * Cycles 5 and 6 of R-CHOP will be administered only to patients with a negative mid-treatment PET scan
  Other Names: Adriamycin ®, Rubex®
Drug: Vincristine — Dose: 1.4 mg/m^2 Administration: IV Push day 1 Schedule: Cycle 1, 2, 3, 4, 5*, 6* (Week 1, 4, 7, 10, 14, 17)
  * Cycles 5 and 6 of R-CHOP will be administered only to patients with a negative mid-treatment PET scan
  Other Names: Oncovin ®, Vincasar Pfs ®, Vincristine Sulfate, LCR, VCR
Drug: Prednisone — Dose: 45 mg/m^2 Administration: IV infusion day 1 (or day 2) over 90 minutes-8 hours Schedule: Cycle 1, 2, 3, 4, 5*, 6* (Week 1, 4, 7, 10, 14, 17)
  * Cycles 5 and 6 of R-CHOP will be administered only to patients with a negative mid-treatment PET scan
  Other Names: Sterapred®, Sterapred® DS, Prednisone Intensol
Drug: Ondansetron — Premedication for R-CHOP Dose: 8 mg Route: PO Schedule: 15 min pre-CHOP chemotherapy
  Other Names: Zofran®, Zofran® ODT, Zuplenz®
Drug: Dexamethasone — Premedication for R-CHOP Dose: 12 mg Route: PO Schedule: 15 min pre-CHOP chemotherapy
  Other Names: Decadron®, Dexamethasone Intensol®, Dexpak® Taperpak®
Drug: Diphenhydramine — Premedication for R-CHOP Dose: 50 mg Route: PO Schedule: Prior to rituximab and then q 4h during rituximab infusion
  Other Names: Aler-Dryl®, Benadryl®, Nytol®, Diphenhist®
Drug: Acetaminophen — Premedication for R-CHOP Dose: 650 mg Route: PO Schedule: Prior to rituximab and then q 4h during rituximab infusion
  Other Names: Tylenol®
Drug: Ifosfamide — R-ICE Chemotherapy Schedule (cycles repeated every 3 weeks) Dose: 5000 mg/m^2 (total dose per cycle) Administration: In 3 equally divided doses IV infusion days 1,2,3, over 2 hours Schedule: Cycle 1, 2, 3, 4 (Week 14, 16, 20, 23)
  Other Names: Ifex®, Isophosphamide
  Arms: R-ICE (Positive Mid-Treatment PET Scan
Drug: Mesna (IV) — R-ICE Chemotherapy Schedule (cycles repeated every 3 weeks) Dose: 5000 mg/m^2 (total dose per cycle) Administration: In 3 equally divided doses IV infusion days 1,2,3 (with ifosfamide) over 2 hours Schedule: Cycle 1, 2, 3, 4 (Week 14, 16, 20, 23)
  Other Names: Mesnex®, Sodium 2-mercaptoethanesulfonate
  Arms: R-ICE (Positive Mid-Treatment PET Scan
Drug: Mesna (oral) — R-ICE Chemotherapy Schedule (cycles repeated every 3 weeks) Dose: 2 g Administration: PO 2h and 4h after ifosfamide infusion on days 1,2,3 Schedule: Cycle 1, 2, 3, 4 (Week 14, 16, 20, 23)
  Other Names: Mesnex®, Sodium 2-mercaptoethanesulfonate
  Arms: R-ICE (Positive Mid-Treatment PET Scan
Drug: Carboplatin — R-ICE Chemotherapy Schedule (cycles repeated every 3 weeks) Dose: 5 x (25+CrCl*) (maximum dose 800 mg) Administration: IV infusion day 1 over 1 hour Schedule: Cycle 1, 2, 3, 4 (Week 14, 16, 20, 23)
  *Carboplatin is dose via the Calvert formula with an AUC of 5, maximum dose 800 mg per cycle.
  Estimate Creatinine Clearance (CrCl)
  Other Names: CBDCA
  Arms: R-ICE (Positive Mid-Treatment PET Scan
Drug: Etoposide — R-ICE Chemotherapy Schedule (cycles repeated every 3 weeks) Dose: 100 mg/m^2 Administration: IV infusion day 1,2,3 over 30 minutes Schedule: Cycle 1, 2, 3, 4 (Week 14, 16, 20, 23)
  Other Names: Etopophos®, VP-16
  Arms: R-ICE (Positive Mid-Treatment PET Scan
Drug: Rituximab — R-ICE Chemotherapy Schedule (cycles repeated every 3 weeks) Dose: 375 mg/m^2 Administration: IV infusion day 1 (or day 2 or day 3) over 90 minutes-8 hours Schedule: Cycle 1, 2, 3, 4 (Week 14, 16, 20, 23)
  Other Names: Rituxan®
  Arms: R-ICE (Positive Mid-Treatment PET Scan
Drug: Ondansetron — Premedication for R-ICE Dose: 8 mg Route: PO Schedule: 15 min pre-chemotherapy daily
  Other Names: Zofran®, Zofran® ODT, Zuplenz®
  Arms: R-ICE (Positive Mid-Treatment PET Scan
Drug: Dexamethasone — Premedication for R-ICE Dose: 8 mg Route: PO Schedule: 15 min pre-chemotherapy daily
  Other Names: Decadron®, Dexamethasone Intensol®, Dexpak® Taperpak®
  Arms: R-ICE (Positive Mid-Treatment PET Scan
Drug: Diphenhydramine — Premedication for R-ICE Dose: 50 mg Route: PO Schedule: Prior to rituximab and then q 4h during rituximab infusion
  Other Names: Aler-Dryl®, Benadryl®, Nytol®, Diphenhist®
  Arms: R-ICE (Positive Mid-Treatment PET Scan
Drug: Acetaminophen — Premedication for R-ICE Dose: 650 mg Route: PO Schedule: Prior to rituximab and then q 4h during rituximab infusion
  Other Names: Tylenol®
  Arms: R-ICE (Positive Mid-Treatment PET Scan
Other: PET Scan — Investigations: 18F-FDG-PET scan Timing: After 4 cycles of R-CHOP (days 21-28) and after 4 cycles of R-ICE (days 28-35)
  Other Names: Positron emission tomography (PET) scan

SUMMARY:
The purpose of this study is to assess whether patients who are likely to fail R-CHOP, as predicted by a mid-treatment PET scan, can have an improved outcome if switched to a standard salvage regimen R-ICE (rituximab, ifosfamide, carboplatin, etoposide).

Patients who have a negative PET scan after 4 cycles of R-CHOP have an excellent prognosis (>85% chance of cure) and should complete treatment with 6 cycles of standard R-CHOP. Patients who have a positive PET scan after 4 cycles of R-CHOP have a very poor prognosis (~10% chance of cure) and may have an improved outcome if switched to a non-cross resistant chemotherapy combination R-ICE.

DETAILED DESCRIPTION:
This is a phase II trial investigating tailoring first-line therapy for advanced stage diffuse large B-cell NHL (DLBCL) based on a mid-treatment 18F-FDG- positron-emission tomography (PET) scan result. More than half of all patients with DLBCL can be cured with 6-8 cycles of standard R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone). Patients who are not cured with R-CHOP have a very poor prognosis. This study will assess whether patients who are likely to fail R-CHOP, as predicted by a mid-treatment PET scan, can have an improved outcome if switched to a standard salvage regimen R-ICE (rituximab, ifosfamide, carboplatin, etoposide).

Objectives:

* To assess the efficacy of tailoring first-line therapy based on a mid- treatment PET scan result for patients with advanced stage DLBCL.
* To assess the progression-free survival (PFS) in patients with advanced stage DLBCL who have a negative mid-treatment PET scan and receive standard therapy with six cycles of CHOP-R and patients with a positive mid-treatment PET scan who receive four cycles of CHOP-R followed by four cycles of R-ICE chemotherapy.
* To assess the overall survival (OS) in patients with advanced stage DLBCL who have a negative mid-treatment PET scan and receive standard therapy with six cycles of CHOP-R and patients with a positive mid-treatment PET scan who receive four cycles of CHOP-R followed by four cycles of R-ICE chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* newly diagnosed histologically proven CD-20 positive diffuse large B- cell lymphoma by tissue biopsy, listed under peripheral B-cell neoplasm according to the WHO/REAL classification (diffuse large B-cell lymphoma, mediastinal large B-cell lymphoma, T-cell rich B-cell lymphoma, intravascular large B-cell lymphoma)
* Advanced stage disease defined as - patients with stage III or stage IV disease; or patients with stage I or stage II disease with one of the following additional criteria: B-symptoms, or disease that is not radio- encompassable within a single involved field, or not a candidate for brief chemotherapy and irradiation, or the presence of bulky disease (any single mass => 10 cm)
* Previously untreated or treated with up to 3 cycles of standard dose 3- weekly R-CHOP chemotherapy prior to enrollment (i.e. patients may be enrolled prior to initiation of the fourth cycle of R-CHOP chemotherapy)
* ECOG Performance Status 0,1 or 2 at time of enrollment
* No evidence of progressive disease while on R-CHOP chemotherapy
* The patient must sign the consent form prior to registration

Exclusion Criteria:

* Patients with a history of any other lymphoproliferative disorder, including prior history of indolent NHL
* Patients with a history of prior or concurrent malignancies within 5 years of the current diagnosis, except adequately treated non- melanoma skin cancer, and curatively treated in-situ cancer of the cervix
* Known HIV infection
* Known hepatitis B virus infection
* Pregnancy or lactation. Men and women of childbearing age must be using adequate contraception.
* Significant renal insufficiency (serum creatinine > 200 mmol/L), unless due to lymphoma
* Significant hepatic insufficiency (serum total bilirubin > 30 mmol/L), unless due to lymphoma
* Cardiac contraindication to doxorubicin therapy (e.g. abnormal contractility on echocardiography). If history of cardiac disease, ejection fraction must be within normal limits for age.
* Neurologic contraindication to vincristine (e.g. peripheral neuropathy)
* Absolute neutrophil count <1.5 x 109/L (unless due to bone marrow involvement with lymphoma or due to initiation of R-CHOP chemotherapy)
* Platelet count < 100 x 109/L (unless due to splenomegaly, bone marrow involvement with lymphoma or due to initiation of R-CHOP chemotherapy)
* Evidence of active systemic infection
* Any medical condition that in the opinion of the investigator would compromise treatment delivery, add toxicity or impair assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-08; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) in participants with advanced stage DLBCL | Estimated two years
  Progression-free survival (PFS) in participants with advanced stage DLBCL who have a negative mid-treatment PET scan and receive standard therapy with six cycles of CHOP-R and patients with a positive mid-treatment PET scan who receive four cycles of CHOP-R followed by four cycles of R-ICE chemotherapy.
  Progression-free survival is defined as the duration of time from diagnosis to time of disease progression or death from any cause. Living patients who have remained free of progression will have their PFS censored on the date last known alive.

SECONDARY OUTCOMES:
Overall survival (OS) in participants with advanced stage DLBCL | Several years
  Overall survival (OS) in participants with advanced stage DLBCL who have a negative mid-treatment PET scan and receive standard therapy with six cycles of CHOP-R and patients with a positive mid-treatment PET scan who receive four cycles of CHOP-R followed by four cycles of R-ICE chemotherapy.
  Overall survival will be defined as the time from diagnosis to the date of death. If the participant is lost to follow-up, survival will be censored on the last date the participant was known to be alive.
The safety of R-ICE therapy in first-line therapy of DLBCL following four cycles of R-CHOP as assessed using the NCI Common Terminology Criteria for Adverse Events Version 3.0 | Six months
Investigate clinical and biologic markers that characterize participant heterogeneity and may serve as predictors of response to therapy and overall outcome. | 1 year
  A central pathology review of original diagnostic biopsies will be performed by pathologists at the Coordinating Center to ensure appropriate lymphoma subclassification. This centralized review is not required prior to enrollment, provided the patients biopsy has been carefully reviewed by local pathologists and determined to be DLBCL.
  Correlative studies of biologic markers will be performed on cases with adequately preserved tissue to explore the biologic heterogeneity between patients and to investigate determinants of response to therapy.
Efficacy of tailoring first-line therapy bases on a mid-treatment PET scan result for patients with advanced stage DLBCL | Four to six months
  All patients will have their BEST RESPONSE on study classified as outlined below. For patients with more than six measurable lesions the six most distinctly measurable at diagnosis should be chosen for response assessment by CT scanning. If available, lesions from both above and below the diaphragm should be chosen, at least two from each region.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie H Sehn, MD, Principal Investigator — BC Cancer Agency - Vancouver Centre
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Jaffe ES, Harris NL, Stein H, Vardiman JW eds. World Health Organization Classification of Tumors. Pathology and Genetics of Tumors of Haematopoietic and Lymphoid Tissues. Lyon: IARC Press; 2001.
- [Background] McKelvey EM, Gottlieb JA, Wilson HE, Haut A, Talley RW, Stephens R, Lane M, Gamble JF, Jones SE, Grozea PN, Gutterman J, Coltman C, Moon TE. Hydroxyldaunomycin (Adriamycin) combination chemotherapy in malignant lymphoma. Cancer. 1976 Oct;38(4):1484-93. doi: 10.1002/1097-0142(197610)38:43.0.co;2-i. PMID 791473
- [Background] Fisher RI, Gaynor ER, Dahlberg S, Oken MM, Grogan TM, Mize EM, Glick JH, Coltman CA Jr, Miller TP. Comparison of a standard regimen (CHOP) with three intensive chemotherapy regimens for advanced non-Hodgkin's lymphoma. N Engl J Med. 1993 Apr 8;328(14):1002-6. doi: 10.1056/NEJM199304083281404. PMID 7680764
- [Background] Anderson DR, Grillo-Lopez A, Varns C, Chambers KS, Hanna N. Targeted anti-cancer therapy using rituximab, a chimaeric anti-CD20 antibody (IDEC-C2B8) in the treatment of non-Hodgkin's B-cell lymphoma. Biochem Soc Trans. 1997 May;25(2):705-8. doi: 10.1042/bst0250705. No abstract available. PMID 9191187
- [Background] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Background] Feugier P, Van Hoof A, Sebban C, Solal-Celigny P, Bouabdallah R, Ferme C, Christian B, Lepage E, Tilly H, Morschhauser F, Gaulard P, Salles G, Bosly A, Gisselbrecht C, Reyes F, Coiffier B. Long-term results of the R-CHOP study in the treatment of elderly patients with diffuse large B-cell lymphoma: a study by the Groupe d'Etude des Lymphomes de l'Adulte. J Clin Oncol. 2005 Jun 20;23(18):4117-26. doi: 10.1200/JCO.2005.09.131. Epub 2005 May 2. PMID 15867204
- [Background] Habermann TM, Weller EA, Morrison VA, et al. Phase III trial of Rituximab-CHOP (R-CHOP) vs. CHOP with a second randomization to maintenance rituximab (MR) or observation in patients 60 years of age and older with diffuse large B-cell lymphoma (DLBCL). Blood. 2003;102:6 abstr.
- [Background] Pfreundschuh M, Trumper L, Gill D, et al. First analysis of the completed Mabthera International (MInT) Trial in young patients with low-risk diffuse large B-cell lymphoma (DLBCL): Addition of rituximab to a CHOP-like regimen significantly improves outcome of all patients with the identification of a very favorable subgroup with IPI=0 and no bulky disease. Blood. 2004;104:48a.
- [Background] Sehn LH, Donaldson J, Chhanabhai M, Fitzgerald C, Gill K, Klasa R, MacPherson N, O'Reilly S, Spinelli JJ, Sutherland J, Wilson KS, Gascoyne RD, Connors JM. Introduction of combined CHOP plus rituximab therapy dramatically improved outcome of diffuse large B-cell lymphoma in British Columbia. J Clin Oncol. 2005 Aug 1;23(22):5027-33. doi: 10.1200/JCO.2005.09.137. Epub 2005 Jun 13. PMID 15955905
- [Background] Philip T, Guglielmi C, Hagenbeek A, Somers R, Van der Lelie H, Bron D, Sonneveld P, Gisselbrecht C, Cahn JY, Harousseau JL, et al. Autologous bone marrow transplantation as compared with salvage chemotherapy in relapses of chemotherapy-sensitive non-Hodgkin's lymphoma. N Engl J Med. 1995 Dec 7;333(23):1540-5. doi: 10.1056/NEJM199512073332305. PMID 7477169
- [Background] Velasquez WS, McLaughlin P, Tucker S, Hagemeister FB, Swan F, Rodriguez MA, Romaguera J, Rubenstein E, Cabanillas F. ESHAP--an effective chemotherapy regimen in refractory and relapsing lymphoma: a 4-year follow-up study. J Clin Oncol. 1994 Jun;12(6):1169-76. doi: 10.1200/JCO.1994.12.6.1169. PMID 8201379
- [Background] Philip T, Armitage JO, Spitzer G, Chauvin F, Jagannath S, Cahn JY, Colombat P, Goldstone AH, Gorin NC, Flesh M, et al. High-dose therapy and autologous bone marrow transplantation after failure of conventional chemotherapy in adults with intermediate-grade or high-grade non-Hodgkin's lymphoma. N Engl J Med. 1987 Jun 11;316(24):1493-8. doi: 10.1056/NEJM198706113162401. PMID 3295541
- [Background] Kewalramani T, Zelenetz AD, Hedrick EE, Donnelly GB, Hunte S, Priovolos AC, Qin J, Lyons NC, Yahalom J, Nimer SD, Moskowitz CH. High-dose chemoradiotherapy and autologous stem cell transplantation for patients with primary refractory aggressive non-Hodgkin lymphoma: an intention-to-treat analysis. Blood. 2000 Oct 1;96(7):2399-404. PMID 11001890
- [Background] Jerusalem G, Beguin Y, Fassotte MF, Najjar F, Paulus P, Rigo P, Fillet G. Whole-body positron emission tomography using 18F-fluorodeoxyglucose for posttreatment evaluation in Hodgkin's disease and non-Hodgkin's lymphoma has higher diagnostic and prognostic value than classical computed tomography scan imaging. Blood. 1999 Jul 15;94(2):429-33. PMID 10397709
- [Background] Hoh CK, Glaspy J, Rosen P, Dahlbom M, Lee SJ, Kunkel L, Hawkin RA, Maddahi J, Phelps ME. Whole-body FDG-PET imaging for staging of Hodgkin's disease and lymphoma. J Nucl Med. 1997 Mar;38(3):343-8. PMID 9074514
- [Background] Carr R, Barrington SF, Madan B, O'Doherty MJ, Saunders CA, van der Walt J, Timothy AR. Detection of lymphoma in bone marrow by whole-body positron emission tomography. Blood. 1998 May 1;91(9):3340-6. PMID 9558391
- [Background] Spaepen K, Stroobants S, Dupont P, Van Steenweghen S, Thomas J, Vandenberghe P, Vanuytsel L, Bormans G, Balzarini J, De Wolf-Peeters C, Mortelmans L, Verhoef G. Prognostic value of positron emission tomography (PET) with fluorine-18 fluorodeoxyglucose ([18F]FDG) after first-line chemotherapy in non-Hodgkin's lymphoma: is [18F]FDG-PET a valid alternative to conventional diagnostic methods? J Clin Oncol. 2001 Jan 15;19(2):414-9. doi: 10.1200/JCO.2001.19.2.414. PMID 11208833
- [Background] Naumann R, Vaic A, Beuthien-Baumann B, Bredow J, Kropp J, Kittner T, Franke WG, Ehninger G. Prognostic value of positron emission tomography in the evaluation of post-treatment residual mass in patients with Hodgkin's disease and non-Hodgkin's lymphoma. Br J Haematol. 2001 Dec;115(4):793-800. doi: 10.1046/j.1365-2141.2001.03147.x. PMID 11843811
- [Background] Zinzani PL, Fanti S, Battista G, Tani M, Castellucci P, Stefoni V, Alinari L, Farsad M, Musuraca G, Gabriele A, Marchi E, Nanni C, Canini R, Monetti N, Baccarani M. Predictive role of positron emission tomography (PET) in the outcome of lymphoma patients. Br J Cancer. 2004 Aug 31;91(5):850-4. doi: 10.1038/sj.bjc.6602040. PMID 15266320
- [Background] Cheson BD, Horning SJ, Coiffier B, Shipp MA, Fisher RI, Connors JM, Lister TA, Vose J, Grillo-Lopez A, Hagenbeek A, Cabanillas F, Klippensten D, Hiddemann W, Castellino R, Harris NL, Armitage JO, Carter W, Hoppe R, Canellos GP. Report of an international workshop to standardize response criteria for non-Hodgkin's lymphomas. NCI Sponsored International Working Group. J Clin Oncol. 1999 Apr;17(4):1244. doi: 10.1200/JCO.1999.17.4.1244. PMID 10561185
- [Background] Juweid ME, Wiseman GA, Vose JM, Ritchie JM, Menda Y, Wooldridge JE, Mottaghy FM, Rohren EM, Blumstein NM, Stolpen A, Link BK, Reske SN, Graham MM, Cheson BD. Response assessment of aggressive non-Hodgkin's lymphoma by integrated International Workshop Criteria and fluorine-18-fluorodeoxyglucose positron emission tomography. J Clin Oncol. 2005 Jul 20;23(21):4652-61. doi: 10.1200/JCO.2005.01.891. Epub 2005 Apr 18. PMID 15837965
- [Background] Spaepen K, Stroobants S, Dupont P, Vandenberghe P, Thomas J, de Groot T, Balzarini J, De Wolf-Peeters C, Mortelmans L, Verhoef G. Early restaging positron emission tomography with ( 18)F-fluorodeoxyglucose predicts outcome in patients with aggressive non-Hodgkin's lymphoma. Ann Oncol. 2002 Sep;13(9):1356-63. doi: 10.1093/annonc/mdf256. PMID 12196360
- [Background] Kostakoglu L, Coleman M, Leonard JP, Kuji I, Zoe H, Goldsmith SJ. PET predicts prognosis after 1 cycle of chemotherapy in aggressive lymphoma and Hodgkin's disease. J Nucl Med. 2002 Aug;43(8):1018-27. PMID 12163626
- [Background] Mikhaeel NG, Timothy AR, O'Doherty MJ, Hain S, Maisey MN. 18-FDG-PET as a prognostic indicator in the treatment of aggressive Non-Hodgkin's Lymphoma-comparison with CT. Leuk Lymphoma. 2000 Nov;39(5-6):543-53. doi: 10.3109/10428190009113384. PMID 11342337
- [Background] Haioun C, Itti E, Rahmouni A, Brice P, Rain JD, Belhadj K, Gaulard P, Garderet L, Lepage E, Reyes F, Meignan M. [18F]fluoro-2-deoxy-D-glucose positron emission tomography (FDG-PET) in aggressive lymphoma: an early prognostic tool for predicting patient outcome. Blood. 2005 Aug 15;106(4):1376-81. doi: 10.1182/blood-2005-01-0272. Epub 2005 Apr 28. PMID 15860666
- [Background] Hutchings M, Mikhaeel NG, Fields P, Nunan T, O'Doherty M, Timothy A. The prognostic value of early FDG-PET during treatment of lymphoma and potential use in response-adapted treatment strategies. Annals of Oncology. 2005;16:280a.
- [Background] Cabanillas F, Hagemeister FB, McLaughlin P, Velasquez WS, Riggs S, Fuller L, Smith T. Results of MIME salvage regimen for recurrent or refractory lymphoma. J Clin Oncol. 1987 Mar;5(3):407-12. doi: 10.1200/JCO.1987.5.3.407. PMID 3819806
- [Background] Velasquez WS, Cabanillas F, Salvador P, McLaughlin P, Fridrik M, Tucker S, Jagannath S, Hagemeister FB, Redman JR, Swan F, et al. Effective salvage therapy for lymphoma with cisplatin in combination with high-dose Ara-C and dexamethasone (DHAP). Blood. 1988 Jan;71(1):117-22. PMID 3334893
- [Background] Moskowitz CH, Bertino JR, Glassman JR, Hedrick EE, Hunte S, Coady-Lyons N, Agus DB, Goy A, Jurcic J, Noy A, O'Brien J, Portlock CS, Straus DS, Childs B, Frank R, Yahalom J, Filippa D, Louie D, Nimer SD, Zelenetz AD. Ifosfamide, carboplatin, and etoposide: a highly effective cytoreduction and peripheral-blood progenitor-cell mobilization regimen for transplant-eligible patients with non-Hodgkin's lymphoma. J Clin Oncol. 1999 Dec;17(12):3776-85. doi: 10.1200/JCO.1999.17.12.3776. PMID 10577849
- [Background] Zelenetz AD, Hamlin P, Kewalramani T, Yahalom J, Nimer S, Moskowitz CH. Ifosfamide, carboplatin, etoposide (ICE)-based second-line chemotherapy for the management of relapsed and refractory aggressive non-Hodgkin's lymphoma. Ann Oncol. 2003;14 Suppl 1:i5-10. doi: 10.1093/annonc/mdg702. PMID 12736224
- [Background] Kewalramani T, Zelenetz AD, Nimer SD, Portlock C, Straus D, Noy A, O'Connor O, Filippa DA, Teruya-Feldstein J, Gencarelli A, Qin J, Waxman A, Yahalom J, Moskowitz CH. Rituximab and ICE as second-line therapy before autologous stem cell transplantation for relapsed or primary refractory diffuse large B-cell lymphoma. Blood. 2004 May 15;103(10):3684-8. doi: 10.1182/blood-2003-11-3911. Epub 2004 Jan 22. PMID 14739217
- [Background] Hertzberg MS, Crombie C, Benson W, Taper J, Gottlieb D, Bradstock KF. Outpatient-based ifosfamide, carboplatin and etoposide (ICE) chemotherapy in transplant-eligible patients with non-Hodgkin's lymphoma and Hodgkin's disease. Ann Oncol. 2003;14 Suppl 1:i11-6. doi: 10.1093/annonc/mdg703. PMID 12736225
- [Background] Vose J, Sneller V. Outpatient regimen rituximab plus ifosfamide, carboplatin and etoposide (R-ICE) for relapsed non-Hodgkin's lymphoma. Ann Oncol. 2003;14 Suppl 1:i17-20. doi: 10.1093/annonc/mdg704. No abstract available. PMID 12736226